CLINICAL TRIAL: NCT04873830
Title: Volumetric Assessment of Volume Stable Collagen Matrix in Soft Tissue Ridge Augmentation At Maxillary Single Implant Site
Brief Title: Volumetric Assessment of Volume Stable Collagen Matrix in Soft Tissue Ridge Augmentation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, ahmed hamdy mahmoud, assistant lecturer of periodontology, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ainshamsUni
Record Dates: First submitted 2021-05-04; First posted 2021-05-05 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Buccal Defect At Implant Sites
Keywords: siebert; dental implant; volume stable collagen matrix; connective tissue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (VCMX) (Experimental): includes 10 patients where implant placement will be performed followed by volume stable collagen matrix placement to augment the buccal defect.
  Interventions: Biological: volume stable collagen matrix placement
- Group II (control) (Experimental): Will include 10 patients where implant placement will be performed followed by connective tissue grafting to augment the buccal defect.
  Interventions: Procedure: connective tissue grafting

INTERVENTIONS:
Biological: volume stable collagen matrix placement — volume stable collagen matrix placement to augment the buccal defect.in class I siebert at the same time of implant placement
  Arms: Group I (VCMX)
Procedure: connective tissue grafting — connective tissue placement to augment the buccal defect.in class I siebert at the same time of implant placement
  Arms: Group II (control)

SUMMARY:
This proposal suggests the use of a collagen scaffold as a core material for GBR in the case of a missing tooth between two existing teeth, in situations where there is sufficient bone to place an implant but a horizontal defect is present in the ridge.

The tested question is whether a thick, reinforced, resorbable collagen scaffold can provide a stable basis for restoring the lost volume of a deficient ridge. As a secondary aim, a positive result could present an option to replace the connective tissue interpositional graft procedure.

DETAILED DESCRIPTION:
• Surgical procedure and clinical measurements:

Pre-surgical phase:

1. Full Conventional non-surgical periodontal therapy involving supra, sub gingival scaling and root planning will be performed
2. Oral hygiene instructions will be repeated until patients had achieved a proper degree of oral hygiene where plaque index (PI) ≤ 1.
3. Four weeks later, patients will be re-evaluated in order to confirm the efficacy of cause related therapy phase.
4. Clinical parameters and CBCT will be recorded prior to surgery.
5. Full arch impressions will be recorded with high viscosity impression material. Baseline casts will be made to be used as a reference for volumetric measurements.

   * Surgical protocol:
   * Patients will undertake implant surgery under local anesthesia for the missing tooth using mid crestal incision at the edentulous area and sulcular incisions at the neighboring mesial and distal teeth.
   * A combined full / partial thickness flap will be made followed by implant placement and healing screw is connected to the implant.
   * For group 1 VCMX will be utilized to graft the buccal defect and primary closure will be achieved using simple interrupted sutures.
   * For group 2 CTG will be utilized to graft the buccal defect and primary closure will be achieved using simple interrupted sutures.
   * Postoperative medications will include (Augmentin 1g twice/day, Flagel 500 mg twice daily and 2 weeks of antiseptic mouth wash ).(Deeb et al , 2015)
   * Patients will be given post-operative instruction and sutures will be removed after 2 weeks.
   * The final abutment will be secured to the implant within 12 weeks after gingival healing for definitive crown placement.

Postoperative surgical evaluation and assessment:

* The follow up period will include oral examination, plaque removal when necessary, at the surgical site.
* Clinical parameters will be measured, impressions redone, and models will be casted 3, 6 and 9 months postoperatively for both groups.
* Radiographic examination using CBCT will be done at 9 months follow up.

Methods of evaluation:

1. Clinical Measurements:

   * Probing depth (Glavind & Loe, 1967).
   * Plaque index (O'leary T, 1972).
   * Bleeding index (Newbrun, 1996)
   * Volumetric changes at the augmented implant site digitally through scanning model casts.

   To assess the volumetric differences between the baseline, 3, 6 and 9 months postoperatively and all the cast models will be transferred to digital replica using an optical scanner. Digital replicas will be produced resembling various time intervals during treatment. Superimposing the different replicas of each case utilizing the best fit algorithm by using reference points from the tooth surfaces. The implant site region will be delineated by the mucogingival line, the mesial and distal papillary midline and the alveolar crest. Thus, any.alterations in volume between the digitized superimposed replicas could be recorded. (Akcali et al., 2015)

   • Pink esthetic score. Pink esthetic score will be recorded for five variables: "mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, and root convexity/soft tissue color and texture at the facial aspect of the implant site". A score of 2, 1, or 0 will be assigned to all five PES parameters.

   The two papillary scores (mesial and distal) will be assessed for the complete presence (score 2), incomplete presence (score 1) or absence (score0) of papillary tissue. The curvature of the facial soft tissue line, also defined as the line of emergence of the implant restoration from the soft tissues, will be evaluated as being identical (score 2 ), slightly different (score 1), or markedly different (score 0) compared to the natural control tooth and thus, provided a natural symmetrical or disharmonious appearance and in comparison to the contralateral tooth in terms of an identical vertical level (score 2), a slight (<1 mm) discrepancy (score 1), or a major (>1 mm) discrepancy (score 0). Finally, the combined three additional specific soft tissue parameters as one variable: the presence, partial presence, or absence of a convex profile (in analogy to a root eminence) on the facial aspect, as-well-as-the-related-mucosal-color-and-surface texture. To achieve a score of 2 for this-combination-variable, all-three-parameters-were more-or-less-identical-compared-to-the-control-tooth. A value of 1 will be given if two criteria are fulfilled, whereas a score of 0 will be given if none or only one parameter matches the control site. (Tettamanti et al, 2014)
   * Visual analogue scale to measure postoperative pain. Pain.score.reported.by.the.patient. directly.through.Visual.Analogue.Scale.score (from 0 to 10. 0: no pain, 1: minimal pain, 5: moderate pain, 10: severe pain) VAS will be recorded after 2 weeks (Yıldırım et al., 2017)
   * The OHIP (OHIP-14 questionnaire) Will be used to assess limitation of function , pain , discomfort, social , psychological ,physical disability and general satisfaction. The OHIP-14 utilizes a scale with five categories (1 = never, 2 = hardly ever, 3 = occasionally, 4 = fairly often, and 5 = very often).A lower score in any of the five categories indicates higher satisfaction. (Al-zubeidi et al, 2011)
   * Soft tissue thickness will be measured at baseline and 9 months postoperatively using.an.anesthetic.needle.with.a.rubber.stopper to pierce the gingiva horizontally and perpendicular to the long axis of the tooth till bone contact 2mm coronal to the MGJ and in the mid distance mesiodistally
   * The part of the instrument penetrating into soft tissue will be measured in mm. (Cairo et al 2017)
2. Radiographic Examination:

   * Cone Beam Computed Tomography (CBCT) will be taken at baseline before implant placement and 9 months later to measure soft tissue thickness.

Statistical analysis:

The collected data will be revised, coded, tabulated and introduced to a PC using Statistical package for Social Science (SPSS 15.0 for windows; SPSS Inc, Chicago, IL, 2001). Data will be presented and suitable analysis will be done according to the type of data obtained for each parameter.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients in a healthy systemic condition.
2. Both genders with age ranging from 20 to 50 years old.
3. Patients should have single missing tooth in anterior or premolar area.
4. Seibert Class I ridge defect.
5. Sufficient bone height and width that doesn't necessitate bone grafting or any other ridge augmentation protocols.
6. Healing period of 3 months after extraction prior to surgical procedures.
7. Patients should approve to deliver a signature to a written consent after study nature explanation.

Exclusion Criteria:

1. Patients with any smoking habits.
2. Pregnant females, decisional impaired individuals, Prisoners and handicapped patients.
3. Patients having poor oral hygiene or not wanting to carry out oral hygiene measures.
4. Patients with infections either periodontally or periapically.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
volumetric changes of soft tissue at implant sites with siebert class I | 9 months
  Is to evaluate the volumetric changes of soft tissues at implant sites with Siebert class I ridge defect after augmentation with volume stable collagen matrix in comparison with connective tissue grafting

SECONDARY OUTCOMES:
esthetic outcome | 9 months
  Pink esthetic score will be recorded for five variables: "mesial papilla, distal papilla, curvature of the facial mucosa, level of the facial mucosa, and root convexity/soft tissue color and texture at the facial aspect of the implant site". A score of 2, 1, or 0 will be assigned to all five PES parameters.
patient satisfaction | 9 months
  using a satisfaction questionnaire

OTHER OUTCOMES:
crestal bone stability | 9 months
  crestal bone level was measured preoperative and 9 months postoperative to check stability of bone level around implant between both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Dental School, Cairo, Egypt